CLINICAL TRIAL: NCT05356429
Title: Study on the Effectiveness of Small Molecule LCDM Combined With Oocyte Activation in Improving GV Oocyte in Vitro Maturation
Brief Title: Small Molecule LCDM and GV Oocyte
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Chen Xi, Associate Researcher, Peking University People's Hospital
Other Study IDs: PKUPHIVF002
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Assisted Reproduction
Keywords: Small molecule LCDM; Oocyte activation; In vitro maturation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental group: In the experimental group, LCDM was added to the general mature culture medium.
  Interventions: Other: Small molecule LCDM
- control group: In the control group, he culture medium was general mature culture medium.

INTERVENTIONS:
Other: Small molecule LCDM — The cocktail of small molecules includes four chemical components of LCDM were added to GV oocyte culture medium.
  Groups: experimental group

SUMMARY:
Immature eggs obtained during the oocyte retrieval cycle are discarded as medical waste because they cannot complete fertilization, but each egg is important for people with poor clinical outcome. In vitro maturation (IVM) technique allows immature GV and MI eggs to mature in vitro, offering hope for this population to increase the clinical pregnancy rate in a single oocyte retrieval cycle. However, the clinical effectiveness of IVM clinical application is still very low, especially the utilization rate of GV eggs is extremely low. The cocktail of small molecules includes four chemical components of LCDM, which are related to cell proliferation, in vitro maturation of eggs, and protection of cells from oxidative stress. Our preliminary experiments confirmed that the addition of a certain concentration of LCDM in the culture medium can significantly improve the in vitro maturation rate and embryo utilization rate of immature GV eggs. In this study, LCDM immature oocyte culture system was used to carry out in vitro maturation culture of GV oocytes, and combined with oocyte activation technology to verify the clinical safety of LCDM in vitro culture system by observing the in vitro maturation rate, fertilization rate and embryo development results of GV oocytes, so as to provide laboratory data for clinical application of GV oocytes in special patients.

ELIGIBILITY:
Inclusion Criteria:

* ICSI cycle with more than 2 GV oocytes

Exclusion Criteria:

* The etiological diagnosis is that the man has extremely severe oligoasthenospermia and primary azoospermia. These patients can lead to low fertilization rate due to sperm, so they are excluded from the group.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: GV oocytes were collected for IVM patients undergoing in vitro fertilization embryo transfer (IVF-ET) in our center. IVM combined with artificial oocyte activity was used to observe and accurately estimate the state of oocyte, then select MII oocyte for the further experiment. All patients in this study were ICSI cycle that the number of oocytes more than two GV oocytes.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of GV oocyte maturation rate at 48 hours | 48 hours
  The GV oocyte maturation rate was defined as the number of MII oocytes which were come from GV oocyte during in vitro maturation. The more MII oocytes, the higher the in vitro maturation rate of the patient's oocytes.
Change from the quality of MII oocytes between the two groups at 48 hours | 48 hours
  The two groups of mature MII eggs were compared, and the chromosome ploidy, spindle integrity and cortical particle distribution were observed respectively to determine the quality of MII eggs in the two groups.
  The evaluation methods include that the chromosomes of normal mature oocytes are aneuploid, the spindles are arranged orderly, and the cortical particles are distributed in the cortical area.